CLINICAL TRIAL: NCT04933695
Title: A Phase 2, Multicenter, Open-label Study of Sotorasib (AMG 510) in Subjects With Stage IV NSCLC Whose Tumors Harbor a KRAS G12C Mutation in Need of First-line Treatment (CodeBreaK 201)
Brief Title: A Study of Sotorasib (AMG 510) in Participants With Stage IV NSCLC Whose Tumors Harbor a KRAS p.G12C Mutation in Need of First-line Treatment
Acronym: CodeBreaK201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190288; 2021-002638-18 (EudraCT Number)
Expanded Access: NCT04667234 (No longer available)
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; KRAS p.G12C; Sotorasib; AMG 510
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotorasib: 960 mg Daily (Experimental): Participants with metastatic non-small cell lung cancer (NSCLC) with Kirsten rat sarcoma (KRAS) p.G12C mutation whose tumors express < 1% programmed death-ligand 1 (PD-L1) and/or serine/threonine kinase 11 (STK11) mutation in need of first line treatment will be administered sotorasib 960 mg daily. Participants will be stratified by known presence of STK11 mutation.
  Interventions: Drug: Sotorasib
- Sotorasib: 240 mg Daily (Experimental): Participants with metastatic non-small cell lung cancer (NSCLC) with Kirsten rat sarcoma (KRAS) p.G12C mutation whose tumors express < 1% programmed death-ligand 1 (PD-L1) and/or serine/threonine kinase 11 (STK11) mutation in need of first line treatment will be administered sotorasib 240 mg daily. Participants will be stratified by known presence of STK11 mutation.
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — Oral tablet
  Other Names: AMG 510; LUMYKRAS; LUMAKRAS

SUMMARY:
The main objective of this study is to evaluate the tumor objective response rate (ORR) assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in participants who receive sotorasib at either 960 mg daily or 240 mg daily whose tumors are programmed death-ligand 1 (PD-L1) Tumor Proportion Score (TPS) < 1% and/or harbor a serine/threonine kinase 11 (STK11) co-mutation, in a subgroup of participants with PD-L1 < 1% and in a subgroup of participants with STK11 co-mutation.

ELIGIBILITY:
Inclusion Criteria:

* Adult (= or > 18 years old) with NSCLC
* Untreated Stage IV metastatic disease. Participants who received adjuvant or neoadjuvant anti-tumor therapy are eligible if the adjuvant/neoadjuvant therapy was completed greater than 12 months prior to the development of metastatic stage IV disease
* Pathologically documented metastatic NSCLC with KRAS G12C mutation (local confirmation)
* Programmed death-ligand 1 (PD-L1) TPS Score < 1% and/or serine/threonine kinase 11 (STK11) co-mutation (local confirmation)
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* No active brain metastases
* Measurable disease per investigator interpretation using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria

Exclusion Criteria:

* Mixed small-cell lung cancer and NSCLC histology
* Myocardial Infarction within 6 months of study Day 1
* Use of proton-pump inhibitors (PPIs), histamine (H2) receptor antagonists (H2RA), strong inducers of cytochrome P450 (CYP) 3A4 (CYP3A4) or known CYP3A4 sensitive substrates or P-gp substrates
* Therapeutic or palliative radiation therapy within 2 weeks of study day 1
* Unable to take oral medication
* Unable to receive both iodinated contrast for computed tomography (CT) scans and gadolinium contrast for magnetic resonance imagine (MRI) scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (OR) | Up to 6 years
  OR is defined as the total of Complete Response (CR) and Partial Response (PR).

SECONDARY OUTCOMES:
Disease Control Rate | Up to 6 years
Duration of Reponse (DOR) | Up to 6 years
Time to Response (TTR) | Up to 6 years
Progression-free Survival (PFS) | Up to 6 years
Overall Survival (OS) | Up to 6 years
Number of Participants with a Treatment-emergent Adverse Event (TEAE) | Day 1 up to Month 13
Number of Participants with a Treatment-related Adverse Event | Day 1 up to Month 13
Number of Participants with a Clinically Significant Change from Baseline in Vital Signs | Baseline (Screening; up to 28 days pre-dose) up to Month 13
Number of Participants with a Clinically Significant Change from Baseline in Electrocardiograms (ECGs) | Baseline (Screening; up to 28 days pre-dose) up to Month 13
Number of Participants with a Clinically Significant Change from Baseline in Clinical Laboratory Tests | Baseline (Screening; up to 28 days pre-dose) up to Month 13
Maximum Plasma Concentration (Cmax) of Sotorasib | Day 1 up to Month 3
Time to Reach Maximum Plasma Concentration (tmax) of Sotorasib | Day 1 up to Month 3
Area Under the Plasma Concentration-time Curve (AUC) of Sotorasib | Day 1 up to Month 3

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (67):
- United States (30):
  - Alabama Oncology, Birmingham, Alabama
  - Arizona Oncology Associates Professional Corporation, Tucson, Arizona
  - City of Hope at Long Beach Elm, Duarte, California
  - City of Hope National Medical Center, Duarte, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Northwest Georgia Oncology Centers PC, Marietta, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Frederick Memorial Hospital, Frederick, Maryland
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at New York University Langone, New York, New York
  - Northport Veterans Affairs Medical Center, Northport, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Duke University Medical Center, Morris Cancer Clinic, Durham, North Carolina
  - Allegheny Health Network Cancer Institute at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Cancer Pavillion, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Plano East, Dallas, Texas
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - Flower Mound, Dallas, Texas
  - Texas Oncology - Baylor, Dallas, Texas
  - Texas Oncology-Denton, Denton, Texas
  - Oncology Consultants PA, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology- Mckinney, McKinney, Texas
  - Texas Oncology - Northeast Texas, Paris, Texas
  - Gundersen Health System, La Crosse, Wisconsin
- Belgium (4):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
- Odense Universitetshospital, Odense C, Denmark
- France (10):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Universitaire Régional de Lille - Hôpital Albert Calmette, Lille
  - Centre Hospitalier Universitaire de Limoges - Hopital Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Montpellier - Val d Aurelle, Montpellier
  - Hopital Cochin, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier de Nantes - Hôpital Nord Laënnec, Saint-Herblain
  - Hôpital Sainte Musse, Toulon
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
- Germany (3):
  - Universitätsklinikum Köln, Cologne
  - Klinikum und Fachbereich Medizin Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main
  - Asklepios - Fachkliniken München-Gauting, Gauting
- Italy (4):
  - Azienda Socio Sanitaria Territoriale di Monza Ospedale San Gerardo, Monza (MB)
  - Azienda Ospedaliera di Rilievo Nazionale Specialistica dei Colli Monaldi, Napoli
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano (TO)
  - Istituti Fisioterapici Ospitalieri Regina Elena San Gallicano, Rome
- Nederlands Kanker Instituut Antoni van Leeuwenhoekziekenhuis, Amsterdam, Netherlands
- Spain (6):
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario La Paz, Madrid
- Sweden (5):
  - Gavle Sjukhus, Gävle
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Universitetssjukhuset i Linkoping, Linköping
  - Skanes Universitetssjukhus, Lund
  - Norrlands Universitetssjukhus, Umeå
- Turkey (Türkiye) (3):
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi, Edirne
  - Koc Universitesi Hastanesi, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com